CLINICAL TRIAL: NCT04451733
Title: Effect of Endotracheal Intubation Performance on the Outcomes in out-of Hospital Cardiac Arrest Patients
Brief Title: Effect of ETI Performance on CPR Outcomes
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Associate Professor, Konkuk University Medical Center
Other Study IDs: INTU_CPRoutcome
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Cardiopulmonary Arrest
Keywords: intubation; Cardiopulmonary Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endotracheal intubation — Perform the endotracheal intubation during CPR

SUMMARY:
This is a clinical observation study based on analysis of video-clip data of cardiopulmonary resuscitation (CPR) for out-of hospital cardiac arrest (OHCA) in emergency department. Aim of study is to evaluate effect of the factors relating endotracheal intubation (ETI) on the outcome of OHCA patients.

DETAILED DESCRIPTION:
ETI is a standard method for placement of advanced airway during CPR. Frequent attempts or delayed ETI may affect adversely on the outcomes of OHCA. However, there was no known detailed data of explaining this issues.

This study tried to evaluate effect of factors of ETI including numbers of trial, time for ETI trial, interruption time and esophageal intubation during CPR on outcomes of OHCA patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffered sudden cardiac arrest and intubated during CPR

Exclusion Criteria:

* case of requesting the do-not-atempt resuscitation
* patients who were diagnosed as adavanced cancer
* cardiac arrest by multiple trauma

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in an urban emergency department at a tertiary hospital in Seoul, Korea
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Good Neurologic outcome | 1 year
  survival with good neurologic status (CPC 1-2) after suffering cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Department of Emergency Medicine, Konkuk University Medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osman AD, Rahman MA, Lam L, Lin CC, Yeoh M, Judkins S, Pratten N, Moran J, Jones D. Cardiopulmonary resuscitation and endotracheal intubation decisions for adults with advance care directive and resuscitation plans in the emergency department. Australas Emerg Care. 2020 Dec;23(4):247-251. doi: 10.1016/j.auec.2020.05.003. Epub 2020 Jun 11. PMID 32534981
- [Background] Panchal AR, Berg KM, Hirsch KG, Kudenchuk PJ, Del Rios M, Cabanas JG, Link MS, Kurz MC, Chan PS, Morley PT, Hazinski MF, Donnino MW. 2019 American Heart Association Focused Update on Advanced Cardiovascular Life Support: Use of Advanced Airways, Vasopressors, and Extracorporeal Cardiopulmonary Resuscitation During Cardiac Arrest: An Update to the American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2019 Dec 10;140(24):e881-e894. doi: 10.1161/CIR.0000000000000732. Epub 2019 Nov 14. PMID 31722552
- [Background] Newell C, Grier S, Soar J. Airway and ventilation management during cardiopulmonary resuscitation and after successful resuscitation. Crit Care. 2018 Aug 15;22(1):190. doi: 10.1186/s13054-018-2121-y. PMID 30111343
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995